CLINICAL TRIAL: NCT00802984
Title: Endovascular Treatment of Thoracic Aortic Aneurysms Using the TALENT Stent Graft System
Brief Title: Endovascular Repair of Descending Thoracic Aortic Aneurysms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-11092007-868; IRB Protocol Number 77836
Record Dates: First submitted 2007-12-04; First posted 2008-12-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

INTERVENTIONS:
Device: Endovascular thoracic aortic aneurysm repair using TALENT TAA Stent Graft System

SUMMARY:
The purpose of this study is to determine whether the system is safe and effective for the intended use of treating descending thoracic aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a candidate for repair of a descending thoracic aortic aneurysm.
2. Patient has one or more of the following:

   * Descending thoracic aneurysm, 5 cm in diameter or greater with proximal and distal neck suitable for stent graft placement.
   * Aneurysm is 4-5 cm in diameter but has increased in size by 0.5 cm in last 6 months.
   * Maximum diameter of aneurysm exceeds one and one-half times the transverse dimension of an adjacent normal aortic segment.
   * Post-traumatic pseudoaneurysm
   * Post-surgical pseudoaneurysm
   * Saccular aneurysm
   * Contained rupture
   * Penetrating ulcer
3. Patient's vascular dimensions must be in the range that can be safely treated with the stent graft and extensions available to the physician at the time of the procedure.
4. Patient has patent iliac or femoral arteries or acceptable retroperitoneal access via the abdominal aorta that allow endovascular access to the aneurysmal site with a 23F delivery catheter, typically used with a 25F introducer sheath
5. Patient has a non-aneurysmal proximal and distal aortic neck diameter between 25 and 36 mm.
6. Patient is American Society of Anesthesiology (ASA) grade 1 through 4.
7. Patient has a stage of disease or condition where there is no comparable or satisfactory alternative device or therapy available for treatment; or the patient has an immediately life-threatening disease in which there is a reasonable likelihood that death will occur within a matter of months or in which premature death is likely without early treatment.
8. Patient is able and willing to comply with 1 month, 6 month, and 1 year follow-up, and willing to comply with annual post-treatment follow-up requirements thereafter.
9. Patient or patient's legal representative understands and has signed an Informed Consent.

Exclusion Criteria:

1. The stent graft would have to be positioned such that there would be no flow to an artery, major branch artery or major branch arteries which supply the spinal cord.
2. The patient has congenital abnormalities in which the placement of the stent graft will cause occlusion of major arterial flow. Such abnormalities should be evaluated prior to treatment.
3. Patient is pregnant.
4. Patient is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta.
5. Patient has connective tissue disease.
6. Patient has a hypercoagulability disorder.
7. Patient is in acute renal failure.
8. Patient has active systemic infection.
9. Patient is less than 18 years old.
10. Patient has less than a one-year life expectancy.
11. Patient is participating in another research study involving an investigational agent for the treatment of Descending Thoracic Aortic Aneurysms.
12. Patient has other medical, social or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
13. Patient is unwilling or unable to return for or comply with follow-up visit schedules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2002-01 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Stent graft migration
Vessel Dissection or perforation
Stent graft occlusion
Collateral vessel occlusion
Aneurysm rupture
Aneurysm exclusion

SECONDARY OUTCOMES:
Technical success
Patency

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Zarins, MD, Principal Investigator — Stanford University; Jason T Lee, MD
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States